CLINICAL TRIAL: NCT07147972
Title: Comparative Study of Nutraceuticals vs. Conventional Prophylactic Therapy in the Management of Migraine
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Kamal Tolba, Associate professor clinical pharmacy department -faculty of pharmacy- fayoum university, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Management of Migraine
Record Dates: First submitted 2025-08-16; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Migraine; Nutraceuticals
Keywords: Migraine; Nutraceuticals
MeSH Terms: conditions — Migraine Disorders | interventions — Propranolol; Magnesium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Conventional Therapy
  Interventions: Drug: Propranolol 80 mg
- Group 2 (Placebo Comparator): Nutraceutical Therapy
  Interventions: Drug: Magnesium 400Mg

INTERVENTIONS:
Drug: Propranolol 80 mg — Propranolol 40-80 mg/day
  Arms: Group 1
Drug: Magnesium 400Mg — Magnesium 400 mg daily
  Arms: Group 2

SUMMARY:
Migraine is a common disabling neurological condition that significantly affects quality of life. While traditional prophylactic treatments (e.g., beta-blockers, antiepileptics) are effective, they may be associated with side effects leading to poor adherence. Recent evidence suggests that nutraceuticals like magnesium, riboflavin, and coenzyme Q10 may provide a safer alternative. This study aims to compare the efficacy and tolerability of these two approaches.

DETAILED DESCRIPTION:
Primary Objective:

- To compare the reduction in the frequency of migraine attacks between patients receiving conventional prophylactic therapy and those receiving a nutraceutical combination.

Secondary Objectives:

* To evaluate changes in migraine intensity (VAS score), duration, and MIDAS score.
* To assess the side effect profile and patient satisfaction with both interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years

  * - Diagnosed with episodic migraine (ICHD-3 criteria)
  * - ≥4 migraine attacks/month for the past 3 months
  * - Willing to provide informed consent

Exclusion Criteria:

* • - Chronic migraine (>15 headache days/month)

  * - Use of other prophylactic treatments in past month
  * - History of secondary headaches
  * - Pregnancy or breastfeeding
  * - Significant renal, hepatic, or cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
migraine intensity using The visual analog scale (VAS score) | 3 months
  To evaluate changes in migraine intensity using the visual analog scale (VAS score) in both groups which is one of the pain rating scales. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm). Normative values are not available. The scale has to be shown to the patient otherwise it is an auditory scale, not a visual one.
migraine duration | 3 months
  To evaluate changes in migraine duration in both groups. The shorter the migraine attack, the better.
MIDAS score (Migraine Disability Assessment) Score | 3 months
  To evaluate changes in MIDAS score (Migraine Disability Assessment) in both groups. Which is a validated, 5-item questionnaire designed to quantify the severity of headache-related disability over the past three months by assessing missed days and reduced productivity in work/school, household chores, and social/family activities. The total score, which can range from 0 to 270, indicates the overall impact of migraines on daily functioning, with higher scores signifying greater disability. MIDAS score. Disability. MIDAS grade ; 0-5. Little or no disability. I ; 6-10. Mild disability. II ; 11-20. Moderate disability.

SECONDARY OUTCOMES:
changes in the frequency of migraine attacks | 3 months
  Number of participants with the change in the frequency of migraine attacks. Less frequency, the better.
side effect profile | 3 months
  To calculate the % of patients who didn't experience side effects of treatment in both interventions using a combination of standardized patient-reported outcome measures (PROMs) like the Treatment Satisfaction Questionnaire for Medication (TSQM) and SATMED-Q, alongside structured side effect symptom scales such as the Numerical Opioid Side Effect (NOSE) survey. I will Collect patient data through self-administered questionnaires and direct interviews, then analyze the frequency, intensity, and impact of adverse effects on daily life to evaluate satisfaction.
patient satisfaction | 3 months
  To calculate the % of patients who were satisfied with the treatment in both interventions using a combination of standardized patient-reported outcome measures (PROMs) like the Treatment Satisfaction Questionnaire for Medication (TSQM) and SATMED-Q, alongside structured side effect symptom scales such as the Numerical Opioid Side Effect (NOSE) survey. I will Collect patient data through self-administered questionnaires and direct interviews, then analyze the frequency, intensity, and impact of adverse effects on daily life to evaluate satisfaction.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charles A. The pathophysiology of migraine: implications for clinical management. Lancet Neurol. 2018 Feb;17(2):174-182. doi: 10.1016/S1474-4422(17)30435-0. Epub 2017 Dec 8. PMID 29229375